CLINICAL TRIAL: NCT05650593
Title: Oral Health Status in a Group of Egyptian Children With Cerebral Palsy: A Cross-sectional Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Khairy Mahmoud, doctor, Cairo University
Other Study IDs: oral health in cp patients
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Cerebral Palsy
Keywords: oral health
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to assess the oral health status in a group of Egyptian children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a group of neuromuscular disorders affecting the development of movement and posture, causing activity limitations. Disturbances to the development of the infant brain may occur early either in utero, during birth or in the first few months of infancy.It may be due to infection, trauma, hypoxia, or hyperbilirubinemia in addition to genetic and biochemical factors. Subsequently, there will be limitations in muscular activity. CP is the most common motor disability occurring during childhood. The prevalence of CP around the world ranges from 1.5 to >4/1000 live births in the developed countries (Al Hashmi et al. 2017).

The CP classification includes four types: spastic, dyskinetic, hypotonic, and mixed, the spastic type being the most common and at times most severe one. Manifestations of cerebral palsy can take on a vast spectrum from minimal symptoms such as minor movement limitation to spasms, muscular rigidity, confinement in a wheelchair, poor bowel control and respiratory problems (Răducanu, Anca et al. 2008).

The patients with cerebral dysfunction may also display mental retardation, epilepsy, sensorial deficiencies (sight and hearing impairment), persistent primitive reflexes, attention-, memory-, learningand emotional problems, language and speaking disturbances (Amit Mani et al. 2015) .

Patients with CP have numerous oral health problems. Neuromuscular disturbances can affect oral health significantly; they may result in changes of the orofacial region's structure and may affect the development of parafunctional habits, including feeding problems, difficulty maintaining oral hygiene (OH), and barriers to oral care access. Malocclusions and tooth wear are common. Experience of dental trauma is also highly prevalent due to instability as a result of neuromuscular defects or seizures (Du et al. 2010).

Children with CP display the same oral pathology as healthy persons. However, they present a higher susceptibility to several oro-dental diseases (dental caries, periodontal disease, dental trauma, malocclusion, bruxism, temporomandibular joint disorders, enamel hypoplasia, abnormal oral habits - tongue thrust, mouth breathing, drooling etc.) due to the abnormal neuromuscular coordination of the tongue, lips, and cheeks and to the low level and the reduced quality of the oral care. The treatment of CP is complex and multidisciplinary, consisting in general (kinetotherapy, surgical interventions, myorelaxants medication) and oral treatment (behavior management, prophylactic, curative) (Sedky 2017).

Parental counselling about diet, oral hygiene procedures and the use of fluorides are preferred to begin as early as possible. Local anaesthesia is not contraindicated; nevertheless sedation is useful to reduce nausea and lingual dystonia, anxiolytic and muscle relaxant drugs such as diazepam are useful as premedication. In some patients, because of uncontrollable movements or poor cooperation, dental treatment has to be carried out under general anaesthesia. Regarding patient access to dental chair, some patients can be treated in their wheelchairs. Preoperative mouthwashes are prevented better administered as a gel or spray) .use of rubber dam and powerful aspiration are needed. The dental chair should be moved slowly to prevent spastic muscle responses (Wasnik et al. 2020).

Also, the oral manifestations of cp are well documented in literature, there have been few studies that actually investigated the prevelance of oral manifestations in cp patients. Thus the aim of the current proposal is to study the prevelance of oral manifestation of cp. (Du et al. 2010).

ELIGIBILITY:
Inclusion Criteria:

Children diagnosed with Cerebral Palsy

• Children aged from 4 to 14years old irrespective of sex.

Exclusion Criteria:

* The child is uncooperative.
* Parents that refused to give informed consent

Ages: 4 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: Egyptian children with cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2022-12-06 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Oral manifestations of cerebral palsy patients | baseline
  assess the oral health status in a group of Egyptian children with cerebral palsy.
  assess the oral health status in a group of Egyptian children with cerebral palsy.
  assess the oral health status in a group of Egyptian children with cerebral palsy.
  assess the oral health status in a group of Egyptian children with cerebral palsy.
  assess the oral health status in a group of Egyptian children with cerebral palsy.
  assess the oral health status in a group of Egyptian children with cerebral palsy.
  assess the oral health status in a group of Egyptian children with cerebral palsy.
  asses Oral manifestations in cerebral palsy patients

CONTACTS AND LOCATIONS:
Overall Officials: cairo university, Principal Investigator — Cairo University
Locations (1):
- The National institute of Neuromotor System in Imbaba, Cairo, Egypt., Cairo, Egypt

REFERENCES:
- [Background] Bensi C, Costacurta M, Docimo R. Oral health in children with cerebral palsy: A systematic review and meta-analysis. Spec Care Dentist. 2020 Sep;40(5):401-411. doi: 10.1111/scd.12506. Epub 2020 Aug 20. PMID 32815638
- [Background] Al-Allaq T, DeBord TK, Liu H, Wang Y, Messadi DV. Oral health status of individuals with cerebral palsy at a nationally recognized rehabilitation center. Spec Care Dentist. 2015 Jan-Feb;35(1):15-21. doi: 10.1111/scd.12071. Epub 2014 Apr 7. PMID 24708141